CLINICAL TRIAL: NCT02693418
Title: A Randomized, Placebo Controlled Pilot Study to Determine the Effect and Duration of Acidform Gel on Vaginal pH
Brief Title: Duration of Effect of Acidform Gel on Vaginal pH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Evofem Inc. (Industry)
Collaborators: Clinical Research Management, Inc. (Industry); Johns Hopkins University (Other); MetroHealth Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EVO-002
Record Dates: First submitted 2016-02-18; First posted 2016-02-26 (Estimated); Results first posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Acidform Gel, Group A (Experimental): Administration of a single vaginal dose of Acidform gel (5 g)
  Interventions: Drug: Acidform 5 g
- Acidform Gel, Group B (Experimental): Administration of a single vaginal dose of Acidform gel (4 g)
  Interventions: Drug: Acidform 4 g
- Acidform Gel, Group C (Experimental): Administration of a single vaginal dose of Acidform gel (3 g)
  Interventions: Drug: Acidform 3 g
- Placebo Gel, Group D (Placebo Comparator): Administration of a single dose of hydroxyethylcellulose (HEC) placebo gel (4 g)
  Interventions: Drug: Placebo 4 g
- No intervention, Group E (No Intervention): No vaginal product administered

INTERVENTIONS:
Drug: Acidform 5 g — Effect of 5 g vaginally administered Acidform on pH over 7 days
  Arms: Acidform Gel, Group A
Drug: Placebo 4 g — Effect of 4 g of vaginally administered HEC placebo gel on pH over 7 days
  Other Names: Natrasol 250 HX Pharm
  Arms: Placebo Gel, Group D
Drug: Acidform 4 g — Effect of 4 g vaginally administered Acidform on pH over 7 days
  Arms: Acidform Gel, Group B
Drug: Acidform 3 g — Effect of 3 g vaginally administered Acidform on pH over 7 days
  Arms: Acidform Gel, Group C

SUMMARY:
The objective of this study was to determine the magnitude and duration of the reduction in pH (acidification) following a single dose of Acidform vaginal gel containing 3, 4, or 5 g compared with hydroxyethylcellulose placebo gel (4 g) or no treatment. Vaginal pH was measured 1 h, 6 h, 12 h, 24 h, then once daily for 7 days. In addition, the participants were assessed for an exploratory endpoint to the determine effect of one dose of Acidform gel (3, 4 or 5 g) or placebo gel (4 g) or no treatment, on asymptomatic bacterial vaginosis (BV).

DETAILED DESCRIPTION:
One hundred healthy volunteer women, 20 per each treatment arm, were treated with either Intravaginal Acidform Gel(IVAG), 5 g dose (GROUP A), Acidform gel, 4 g dose (GROUP B), Acidform gel, 3 g dose (GROUP C), Universal Placebo Gel (UPG), 4 g (GROUP D) or no treatment (GROUP E). For GROUPS A, B, C and D, treatment is defined as speculum exam plus instillation of Investigational Product (IP) or placebo gel. For GROUP E (control), no treatment is defined as speculum exam and no gel instillation.

At least 15 women in each group were of either African American or Hispanic ethnicity. Routine screening tests were performed on admission; and subjects assessed for BV via vaginal swabs obtained for grading by Amsel criteria.

A direct vaginal pH reading by research staff- was obtained before the speculum exam, as well as one hour, and six hours post-treatment (Day 0). At the one hour and six hour post treatment time points, the direct vaginal pH readings were taken on specimens collected from two different positions in the vagina, in case of incomplete distribution of the IP soon after administration. Both readings are included as data points. At the six hour timepoint, subjects were trained on self-collecting vaginal swabs and performing the vaginal pH test. At 12 hours post-treatment, subjects performed the vaginal pH test themselves using self-obtained swabs, and record their results for clinician review.

Subjects stayed overnight in the domiciliary unit, and vaginal pH and Amsel criteria was measured again by research staff at 24 (+/- 2) hours post-treatment before discharge on Day 1. The subjects were discharged with the appropriate pH testing supplies and diary. All women agreed to abstain from sexual intercourse, douching and use of any intravaginally applied products or devices until after their final study visit on Day 7.

Subjects measured their vaginal pH at 24 (+/-2) hour intervals for 5 days (Days 2-6) as outpatients and recorded the pH test results, and any change in vaginal comfort, in a provided diary. Subjects also recorded any activities engaged in from the abstinence criteria in the study exclusion list, if applicable, each day. On Day 7, subjects returned to the clinic with their diaries, had their vaginal pH and Amsel criteria determined by the clinic staff, and queried as to any vaginal discomfort (vaginal comfort assessment) over the course of the study, as self-recorded in their diaries.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female subjects between 18 and 45 years, inclusive
2. Ability to understand the consent process and procedures
3. Subjects agree to be available for all study visits
4. Written informed consent in accordance with institutional guidelines
5. Negative pregnancy test
6. Able and willing to comply with all study procedures
7. Have not engaged in sexual intercourse, douching or used of any form of vaginal suppository or intravaginal device for 24 hours prior to enrollment.
8. Agree to abstain from sexual intercourse, douching or any form of vaginal suppository or intravaginal device use during course of study
9. Report menstrual cycle regularity (25- to 35- day menstrual cycles)

Exclusion Criteria:

1. Participation in any study with an investigational compound or device within 30 days prior to signing informed consent
2. Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study protocol
3. Any other medical condition(s) that, in the judgment of the investigator, might interfere with the study or require treatment that might interfere with the study
4. Family member of the investigation study staff
5. Pregnant or breast-feeding
6. Inability to provide informed consent
7. A subject with a history or expectation of noncompliance with medications or treatment protocol
8. Women with symptoms of Urinary Tract Infection (UTI) or Sexually Transmitted Infection (STI) reported or observed during examination, at screening*.
9. Women who regularly use douches, vaginal medications or suppositories, feminine sprays, genital wipes or contraceptive spermicides, or report abnormal vaginal discharge in the past 48 hours prior to screening
10. Women who are menstruating or who would expect to menstruate during the study
11. Women who are currently using contraceptives that are directly delivered to the vaginal mucosa, such as NuvaRing
12. Any specific condition that, in the judgment of the Investigator, precludes participation because it could affect subject safety

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2016-08-24 (Actual); Primary Completion 2016-12-12 (Actual); Study Completion 2016-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Avery, MD, Principal Investigator — Metro Health Medical Center; Seema Nayak, MD, Principal Investigator — Johns Hopkins University; John M Griffiss, MD, Study Director — Clinical Research Management, Inc.
Locations (2):
- United States (2):
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Metro Health Medical Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acidform Gel, Group A | Acidform Gel, Group B | Acidform Gel, Group C | Placebo Gel, Group D | No Intervention, Group E
Started | 22 | 21 | 21 | 20 | 21
Completed | 21 | 19 | 19 | 20 | 21
Not Completed | 1 | 2 | 2 | 0 | 0
Not completed — Lost to Follow-up | 1 | 2 | 0 | 0 | 0
Not completed — Menses during study period | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Total: Total of all reporting groups
Arm/Group | Acidform Gel, Group A | Acidform Gel, Group B | Acidform Gel, Group C | Placebo Gel, Group D | No Intervention, Group E | Total
Number analyzed (Participants) | 22 | 21 | 21 | 20 | 21 | 105
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.62 (7.11) | 28.57 (7.20) | 28.12 (5.40) | 30.42 (6.47) | 30.21 (6.45) | 29.8 (6.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 21 | 20 | 21 | 105
  Male | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 2 | 6 | 3 | 23
  Not Hispanic or Latino | 16 | 15 | 19 | 14 | 18 | 82
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 10 | 11 | 8 | 6 | 12 | 47
  White | 10 | 6 | 11 | 11 | 7 | 45
  More than one race | 1 | 4 | 1 | 3 | 1 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: pounds] — Population: One subject in the IVAG acid form 3g group had missing weight data.
  pounds
    number analyzed (Participants) | 22 | 21 | 20 | 20 | 21 | 104
    (all) | 169.54 (49.56) | 169.85 (41.48) | 183.81 (52.97) | 171.40 (42.27) | 177.09 (48.91) | 174.23 (46.65)
Height [Mean (Standard Deviation); unit: Inches] — Population: One subject in the IVAG acid form 3g group had missing height data
  Inches
    number analyzed (Participants) | 22 | 21 | 20 | 20 | 21 | 104
    (all) | 65.19 (2.55) | 64.62 (2.27) | 63.74 (2.89) | 63.91 (2.47) | 64.77 (2.62) | 64.46 (2.57)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: One subject in the IVAG acid form 3g group did not have BMI data
  kg/m^2
    number analyzed (Participants) | 22 | 21 | 20 | 20 | 21 | 104
    (all) | 28.02 (7.55) | 28.59 (6.69) | 31.87 (9.30) | 29.84 (8.51) | 29.55 (7.13) | 29.53 (7.82)

OUTCOME MEASURES:

1. Primary Outcome: Change in Vaginal pH Following a Single Dose of Acidform (3, 4, and 5 g), HEC Placebo (4 g), or no Intervention.
Description: Vaginal swabs were used to collect samples from the vagina of women dosed with Acidform, HEC placebo, or no treatment. The pH of the samples was measured at pre-determined time points over the course of 7 days.
Time Frame: Baseline (Day 0), 1, 6 & 12 hours post treatment, and Days 1, 2, 3, 4, 5, 6 & 7.
Population: Summary of Changes from Baseline (baseline value for vaginal pH is the Pre-Dose measurement on Day 0). Vaginal pH was obtained by the subject on Day 0 (12 hours post treatment only), Day 2, Day 3, Day 4, Day 5 and Day 6. All other vaginal pH values were obtained by the Research staff.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Acidform Gel, Group A | Acidform Gel, Group B | Acidform Gel, Group C | Placebo Gel, Group D | No Intervention, Group E
Number analyzed (Participants) | 22 | 21 | 21 | 20 | 21
pH
  Baseline measure (Day 0) | 4.85 (0.55) | 4.81 (0.62) | 4.91 (0.57) | 5.00 (.069) | 4.77 (0.60)
  1 hour Post-Tx Summary of Changes from Baseline | -0.44 (0.50) | -0.19 (0.54) | -0.30 (0.66) | -.031 (0.55) | -0.16 (0.45)
  6 hour Post-Tx Summary of Changes from Baseline | -0.59 (0.50) | -0.51 (0.57) | -0.49 (0.47) | -0.16 (0.53) | -0.02 (0.50)
  12 hour Post-tx Summary Changes from baseline: number analyzed (Participants) | 21 | 20 | 21 | 20 | 21
  12 hour Post-tx Summary Changes from baseline | -0.76 (0.57) | -0.72 (0.57) | -0.58 (0.70) | -0.02 (0.55) | 0.01 (0.34)
  Day 1 Summary of Changes from Baseline: number analyzed (Participants) | 21 | 20 | 21 | 20 | 20
  Day 1 Summary of Changes from Baseline | -0.72 (0.55) | -0.50 (0.54) | -0.29 (0.65) | -0.13 (0.35) | 0.19 (0.64)
  Day 2 Summary of Changes from Baseline: number analyzed (Participants) | 21 | 19 | 20 | 20 | 21
  Day 2 Summary of Changes from Baseline | -0.33 (0.42) | -0.43 (0.42) | -0.25 (0.39) | 0.23 (0.65) | -0.01 (0.43)
  Day 3 Summary of Changes from Baseline: number analyzed (Participants) | 21 | 19 | 20 | 20 | 21
  Day 3 Summary of Changes from Baseline | -0.40 (0.43) | -0.34 (0.56) | -0.10 (0.50) | 0.05 (0.64) | 0.04 (0.47)
  Day 4 Summary of Changes from Baseline: number analyzed (Participants) | 21 | 19 | 20 | 20 | 21
  Day 4 Summary of Changes from Baseline | -0.38 (0.46) | -0.34 (0.39) | -0.22 (0.47) | 0.11 (0.68) | 0.06 (0.37)
  Day 5 Summary of Changes from Baseline: number analyzed (Participants) | 21 | 19 | 20 | 20 | 21
  Day 5 Summary of Changes from Baseline | -0.36 (0.44) | -0.24 (0.52) | -0.25 (0.36) | -0.25 (0.43) | 0.09 (0.58)
  Day 6 Summary of Changes from Baseline: number analyzed (Participants) | 19 | 19 | 17 | 19 | 20
  Day 6 Summary of Changes from Baseline | -0.46 (0.51) | -0.18 (0.77) | -0.24 (0.49) | -0.19 (0.47) | -0.01 (0.62)
  Day 7 Summary of Changes from Baseline: number analyzed (Participants) | 20 | 19 | 19 | 20 | 21
  Day 7 Summary of Changes from Baseline | -0.14 (0.50) | -0.16 (0.48) | -0.19 (0.48) | -0.16 (0.64) | -0.06 (0.52)

2. Other Pre Specified Outcome: The Effect of a Single Dose of Acidform Gel (3, 4 or 5 g), Placebo Gel (4 g), or no Treatment on Asymptomatic Bacterial Vaginosis (BV) Based on Amsel Criteria.
Description: Amsel Criteria was used at baseline (day 0), compared to Day1 and Day 7 following the single dose of Acidform or placebo. Amsel criteria assessments consisted of Yes/No indications for the presence of each of the following: Vaginal pH> 4.5; Presence of thin, grayish white vaginal discharge; Positive wet prep; Positive whiff amine test. Based on the individual criteria, a derived overall result (positive/negative) was reported. Amsel Result was automatically calculated based whether or not subject is positive in three of the four criteria listed above.
Time Frame: Baseline (Day 0), Day 1 and Day 7
Population: Day 0 (Baseline), Day 1 and Day 7, Amsel Tests Overall results
Measure: Count of Participants; unit: Participants
Arm/Group | Acidform Gel, Group A | Acidform Gel, Group B | Acidform Gel, Group C | Placebo Gel, Group D | No Intervention, Group E
Number analyzed (Participants) | 22 | 21 | 21 | 20 | 21
Participants
  Baseline Day 0 Positive | 4 | 2 | 1 | 4 | 1
  Baseline Day 0 Negative | 18 | 19 | 20 | 16 | 20
  Day 1 Positive: number analyzed (Participants) | 20 | 20 | 20 | 19 | 20
  Day 1 Positive | 0 | 2 | 1 | 1 | 3
  Day 1 Negative: number analyzed (Participants) | 20 | 20 | 20 | 19 | 20
  Day 1 Negative | 20 | 18 | 19 | 18 | 17
  Day 7 Positive: number analyzed (Participants) | 19 | 18 | 17 | 20 | 21
  Day 7 Positive | 1 | 2 | 1 | 2 | 1
  Day 7 Negative: number analyzed (Participants) | 19 | 18 | 17 | 20 | 21
  Day 7 Negative | 18 | 16 | 16 | 18 | 20

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Acidform Gel, Group A | Acidform Gel, Group B | Acidform Gel, Group C | Placebo Gel, Group D | No Intervention, Group E
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/21 | 0/21 | 0/20 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21 | 0/21 | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 16/22 | 13/21 | 16/21 | 13/20 | 10/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acidform Gel, Group A (N=22) | Acidform Gel, Group B (N=21) | Acidform Gel, Group C (N=21) | Placebo Gel, Group D (N=20) | No Intervention, Group E (N=21)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical discharge (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 3 (3)
Cervix disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Cervix inflamation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 15 (19) | 13 (19) | 12 (18) | 10 (14) | 3 (4)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Vaginal odour (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vulvovaginal pain (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 3 (3) | 2 (3) | 1 (1) | 3 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
Low number of subjects at each time point and lost specimens meant a complete analyses were not conducted on specimens from all subjects at all time points and further studies are required to confirm these findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less